CLINICAL TRIAL: NCT01942616
Title: Media, Public Health, and Colluding With Murder: The Development of a Domestic Violence Perpetrator Collusion Measurement Tool.
Brief Title: The Development of a Domestic Violence Perpetrator Collusion Measurement Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: 0910005885
Record Dates: First submitted 2013-08-30; First posted 2013-09-16 (Estimated); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Intimate Partner Violence (IPV)
Keywords: IPV

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Condition 1 (Experimental): Each study arm contains different scenarios presented to the participant.
  Condition 1 is a Perpetrator Positive scenario.
  The content of the Condition 1 group is as follows:
  Framing: Episodic Labeling: DV label Extraneous Information: Perpetrator positive non relevant Victim/Perp Characteristic: Negative victim
  Interventions: Other: Condition 1: Perpetrator Positive
- Condition 2 (Experimental): Each study arm contains different scenarios presented to the participant.
  Condition 2 is a Perpetrator Negative scenario.
  The content of the Condition 2 group is as follows:
  Framing: Thematic Labeling: Assault label Extraneous Information: Perpetrator neutral non relevant Victim/Perp Characteristic: Negative Perpetrator
  Interventions: Other: Condition 2: Perpetrator Negative
- Condition 3 (Placebo Comparator): Each study arm contains different scenarios presented to the participant.
  The content of the Condition 3 group is as follows:
  Framing: Neither Labeling: No label Extraneous Information: None Victim/Perp Characteristic: None
  Interventions: Other: Condition 3: Placebo

INTERVENTIONS:
Other: Condition 1: Perpetrator Positive — Condition 1 frames the event as episodic, labels the event as domestic violence, uses a positive description of the perpetrator, and a negative description of the victim.
  Arms: Condition 1
Other: Condition 2: Perpetrator Negative — The condition 2 intervention/exposure frames the event as thematic, labels the event as assault, uses a neutral description of the perpetrator, and a negative description of the perpetrator.
  Arms: Condition 2
Other: Condition 3: Placebo — This intervention provides no details for the participant and is for comparison use in the study.
  Arms: Condition 3

SUMMARY:
We propose an experimental design to empirically establish the potential link between the media portrayal of DV and changes in an individual's DV descriptive and injunctive social norms. Specifically, this study will measure the degree to which people implicitly collude with DV perpetration.

DETAILED DESCRIPTION:
Aim 1: To determine the impact of media "frames," "labeling," and "information inclusion" on "implicit collusion" with a DV perpetrator.

Hypotheses: Consumers exposed to media reports using "thematic frames" will be less likely to implicitly collude with perpetrators than those exposed to "episodic frames." Consumers exposed to DVH news stories labeled as "domestic violence" will be less likely to implicitly collude with perpetrators than consumers exposed to news stories labeled as "assault." Implicit collusion will correlate positively with the addition of non-relevant perpetrator "humanizing" characteristics. Consumers given negative information about the victim of DVH will be more likely to implicitly collude with the perpetrator than consumers given negative information about the perpetrator.

Aim 2: To determine how media portrayals of domestic violence impact descriptive and injunctive norms about domestic violence and, ultimately, drive implicit collusion with perpetrators.

Hypotheses: Controlling for individual pre-existing attitudes and social norms, consumers exposed to thematic frames or the label of DV will be less likely to shift their norms in a way that supports DV than those exposed to episodic frames or the label of assault. Consumers provided negative victim information or non-relevant characteristics that humanize the perpetrator will be more likely to shift their norms to accept DV.

Exploratory Aim: To identify racial/ethnic, gender, age, and regional differences in DV social norms.

Hypothesis: The media will differentially impact subpopulation DV attitudes, social norms and implicit collusion.

ELIGIBILITY:
Inclusion Criteria:

* Members of the public who are 18 years or older, who identify as White or African American or Hispanic.

Exclusion Criteria:

* Members of the public will be excluded if they are unable to read or understand English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline on The Collusion Framing Subscale | The scale is administered at baseline and then following the sub experiment for a total of 2 times, 30 minutes apart.
  The scale will be developed based on the changes from baseline.
Change from Baseline on The Collusion Labeling Subscale | The scale is administered at baseline and then following the sub experiment for a total of 2 times, 30 minutes apart.
  The scale will be developed based on the changes from baseline.
Change from Baseline on The Collusion Extraneous Information Subscale | The scale is administered at baseline and then following the sub experiment for a total of 2 times, 30 minutes apart.
  The scale will be developed based on the changes from baseline.
Change from Baseline on The Collusion Negative Characteristics Subscale | The scale is administered at baseline and then following the sub experiment for a total of 2 times, 30 minutes apart.
  The scale will be developed based on the changes from baseline.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Yale University, New Haven, Connecticut
  - Loyola University New Orleans, New Orleans, Louisiana
  - Michigan State University, East Lansing, Michigan
  - Michigan Department of Community Health, Lansing, Michigan